CLINICAL TRIAL: NCT00836290
Title: Positive Lifestyles Using Safety
Acronym: Project PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH); Yale AIDS Program (Unknown); AIDS Project Hartford (Industry); Connecticut State, Department of Correction (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 0701002257; UR6PS000391 (NIH)
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: HIV; HIV Infections
Keywords: risk reduction; HIV prevention; HIV education; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-release (Experimental): Participants in the pre-release intervention group will receive four sessions in the four-week period prior to release and will receive a comprehensive booster session four weeks after release.
  Interventions: Behavioral: Pre-Release (Group 1)
- Post-release (Experimental): Participants in the post-release intervention group will receive one comprehensive introductory session four weeks before release and four sessions during the four-week period after release.
  Interventions: Behavioral: Post-release (Group 2)
- Control (No Intervention): Participants in the control group do not receive education sessions during their term in the study. However, these sessions are available to them after completing the study.

INTERVENTIONS:
Behavioral: Pre-Release (Group 1) — Participants in the pre-release intervention group will receive four sessions in the four-week period prior to release and will receive a comprehensive booster session four weeks after release.
  Arms: Pre-release
Behavioral: Post-release (Group 2) — Participants in the post-release intervention group will receive one comprehensive introductory session four weeks before release and four sessions during the four-week period after release.
  Arms: Post-release

SUMMARY:
Project PLUS tests an HIV risk reduction/adherence behavioral intervention with HIV-infected individuals in Connecticut prisons. Participants are randomly assigned to one of three groups: prior to release from incarceration (Group 1), after release from incarceration (Group 2), and treatment-as-usual (Group 3). We hypothesize that the intervention groups (Groups 1 & 2) will demonstrate significantly greater knowledge regarding drug- and sex- related HIV risk behavior and HIV medication adherence, greater motivation to reduce HIV risk behavior and improve HIV medication adherence, and enhanced skills for engaging in HIV risk reduction behavior and HIV medication adherence vs. the treatment-as-usual group. We will also compare these outcomes between Groups 1 and 2.

DETAILED DESCRIPTION:
Project PLUS is an HIV risk reduction/Highly Active Antiretroviral Therapy (HAART) adherence behavioral intervention for persons being released from prisons in Connecticut. The intervention is delivered one-on-one to HIV-infected individuals prior to release from incarceration (Group 1) vs. after release from incarceration (Group 2) vs. treatment as usual (Group 3). The primary hypothesis is that the intervention groups (Groups 1 & 2) will demonstrate significantly greater reduction in rates of HIV sexual and drug risk behaviors and a significantly greater increase in HAART adherence compared to Group 3 participants at 4 months following release from prison. (However, those in Group 3 may come back to participate in the educational sessions, as non-study participants, after their participation has been completed). Based on the IMB model of health behavior change, the primary outcomes of interest are HIV risk reduction knowledge, motivation, behavioral skills (Fisher & Fisher, 1992) and specific event-level partner-by-partner drug and sex risk outcomes including the frequency of unprotected sex episodes across different partners categorized by perceived HIV-status of each partner, numbers of different sexual partners, changes in the frequency of condom use, changes in reported adherence to HIV medication, and changes in reported drug use episodes across different partners categorized by perceived HIV-status of each partner. Additional outcomes of interest include greater knowledge regarding drug- and sex- related HIV risk behaviors and HAART adherence, greater motivation to reduce HIV risk behaviors and improve HAART adherence, enhanced skills for engaging in HIV risk reduction behaviors and HAART adherence. A comparison between Groups 1 & 2 has never been examined, so an important part of this study is to explore this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Meet DSM-IV criteria for opioid-dependence
* Are scheduled to be released from prison within the next 30 days
* Are confirmed to be HIV-infected
* Report drug- or sex-related HIV risk behavior prior to incarceration
* Are willing to provide locator information
* Able to read and understand the questionnaires and consent form
* No minimum duration of incarceration
* Available for the full duration of the study with no anticipated circumstances impeding participation (e.g., pending court case or warrant).

Exclusion Criteria:

* Have an untreated bipolar or psychotic disorder
* Suicidal or homicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected sex episodes across different partners categorized by perceived HIV-status of each partner | Pre-release, Day of Release, 1-mo ff-up, 3-mo ff-up
Numbers of different sexual partners | Pre-release, Day of Release, 1-mo ff-up, 3-mo ff-up
Changes in the frequency of condom use reported | Pre-release, Day of Release, 1-mo ff-up, 3-mo ff-up
Changes in reported HIV medication adherence | Pre-release, Day of Release, 1-mo ff-up, 3-mo ff-up
Changes in reported drug use episodes across different partners categorized by perceived HIV-status of each partner | Pre-release, Day of Release, 1-mo ff-up, 3-mo ff-up

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University
Locations (1):
- Yale AIDS Program, Yale University School of Medicine, New Haven, Connecticut, United States